CLINICAL TRIAL: NCT03565380
Title: Acceptability and Feasibility of a Community-based Strength, Balance and Tai Chi Rehabilitation Program in Improving Physical Function and Balance of Patients After Total Knee Arthroplasty: a Pilot Randomized Controlled Trial
Brief Title: Effectiveness of a Community-based Multi-modal Tai Chi Rehabilitation Program for Patients After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20171225001AW
Record Dates: First submitted 2018-05-30; First posted 2018-06-21 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Total Knee Arthroplasty
Keywords: Tai Chi; Lower limb muscle strength; Balance; Rehabilitation; Multi-faceted intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The reassessments at 6-, 12-, 24-, and 52 weeks, and prospective falls evaluation will be conducted by assessors blinded to group allocation. Due to the nature of the trial, the certified Tai Chi instructor who provides treatments and participants will not be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with intervention (Experimental): 12-week community-based Tai Chi rehabilitation program starting at 12 weeks after TKA
  Interventions: Other: 12-week community-based multi-model Tai Chi rehabilitation program
- Patients without intervention (Experimental): usual post-operative care
  Interventions: Other: Usual post-operative care
- Asymptomatic controls (Experimental): untreated asymptomatic controls
  Interventions: Other: Untreated asymptomatic controls

INTERVENTIONS:
Other: 12-week community-based multi-model Tai Chi rehabilitation program — Participants will receive 12 x 90 minute sessions of supervised exercises over 12 weeks. In addition to usual care, supervised exercise will be held at the Center of Sports Training and Rehabilitation inside the University and each class will be restricted to no more than 8 participants to ensure sufficient personalized attention. Each training session involves warm-up together with stretching of lower extremity muscles, strengthening exercises of the major lower extremity muscle groups by Theraband, balancing exercise, Tai Chi training, and rest/ cool-down. All lower-extremity exercises will be performed bilaterally.
  Other Names: Fall prevention program
  Arms: Patients with intervention
Other: Usual post-operative care — No intervention will be provided
  Arms: Patients without intervention
Other: Untreated asymptomatic controls — No intervention will be provided
  Arms: Asymptomatic controls

SUMMARY:
The rate of falls in patients after total knee arthroplasty (TKA) is high and related to lower limb muscle weakness and poor balance control. However, since routine post-TKA rehabilitation is uncommon, it is paramount to explore alternative strategies to enhance balance and physical functioning in post-TKA patients. As Tai Chi is a proven strategy for improving balance in older people, the proposed study aims to determine the feasibility and acceptability of a 12-week community-based post-TKA multimodal Tai Chi program and to collect preliminary data with respect to the efficacy of such a program in improving balance and physical functioning in post-TKA patients as compared to usual postoperative care.

DETAILED DESCRIPTION:
This is a single-blinded 2-arm RCT. TKA participants will be randomized to either a 12-week community-based rehabilitation program starting at 12 weeks after TKA, or usual post-operative care without outpatient physiotherapy. A third group of asymptomatic controls will be recruited to provide comparisons at various time points. All post-TKA participants will undergo five clinical assessments: 1 week before TKA, and at 6, 12, 24 and 52 weeks after TKA. The untreated asymptomatic controls will be assessed at baseline, and 12 and 52 weeks from baseline

ELIGIBILITY:
Inclusion Criteria:

1. 60 years or above;
2. candidates for primary unilateral TKA who are placed on the TKA waiting list for less than 1 month before their surgery;
3. living independently in the community

Exclusion Criteria:

1. living in assisted living facilities, requiring nursing care, or planning to reside away from the hospital district within 1 year.
2. unstable medical conditions,
3. fracture of lower limbs,
4. malignancy in the last five years,
5. lower limb prosthesis/amputation,
6. congenital defect that is considered to cause the present complaint,
7. systemic inflammatory and autoimmune diseases,
8. previous osteotomy,
9. neurological diseases (e.g. Parkinson's disease, stroke),
10. blindness, revision TKA,
11. complications after primary TKA,
12. cognitive impairment with a Mini-Mental State Examination score < 19
13. prior experience in practicing Tai Chi exercise for at least 3 months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-11-11 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of recruitment and rate of retention | After 52 week post-TKA follow-up
  The recruitment and attrition rates will be monitored on a monthly basis to determine the presence of any specific trends. The recruitment rate (all potential participants), retention and attrition rates (all randomized participants) and completion rates (all enrolled participants) will be assessed at the end of study. Reasons for ineligibility, and/or non-recruitment of eligible patients will be recorded and grouped into categories.
Facilitators and barriers of the intervention | During the intervention and after 52 week post-TKA follow-up
  Attendance and exercise logbooks will be used to monitor non-adherence. The instructor will communicate with non-adherent participants to understand the reasons and barriers for non-adherence and to develop appropriate strategies to improve adherence. Furthermore, to assess the acceptability of the intervention, each participant in the intervention group will be invited to participate in a face-to-face or video call interviews semi-structured interview based on participants' preferences within 1 month after the final follow-up.
Sample size estimation for the future definitive trial | After 52 week post-TKA follow-up
  Based on the standard deviation (SD) of The Chinese version of the Knee Injury and Osteoarthritis Outcome Scale (the higher the score, the better the performance )so as to inform the sample size calculation for the effectiveness trial.
Self-reported physical function | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  The Chinese version of Knee Injury and Osteoarthritis Outcome Scale will be used to document self-reported physical function and to evaluate knee status before/after TKA
Number of trips/falls | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  The number of trips, falls and fall-related injuries in the 12 months before baseline will be documented.

SECONDARY OUTCOMES:
Objective measures of static and dynamic stability | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  When wearing the sensors, participants will perform a tandem stance test with eyes open and eyes closed, the TUG and the 6MWT.
Knee pain | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  It will be measured by an 11-point numeric pain rating scale, which ranges from 0 (no pain) to 10 (the worst imaginable pain). It documents the current, best, and worst pain in the last 24 hours. It will be used to record the pain intensity of participant's knee and other body parts, if appropriate.
Depression | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  Depressive symptoms will be examined by the short form Chinese version of the Geriatric Depression Scale, which comprises 15 questions.
Physical activity level | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  Physical activity will be assessed by the Physical Activity Scale for the Elderly (Chinese version), which is a 12-item questionnaire that documents leisure, physical, household and work-related activities over the last 7 days.
Fear of falling | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  Concern of falling will be measured with the Falls Efficacy Scale, which showed good reliability and validity in measuring fear of falling in frail older people.
Global impression of change | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  Symptom severity, treatment response and the efficacy of treatment 24-weeks post-TKA will be measured by the Global Impression of change scale.
Joint range of motion | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  The ranges of motion of hip, knee, and ankle joints will be evaluated using a goniometer. These assessments are chosen because limited knee/ankle joint ranges have been reported as potential risk factors for falls.
Balance assessment | 1-week before TKA, 6-, 12-, 24- and 52-week post-TKA follow-ups
  The Brief-Balance Evaluation Systems test comprises six static and six dynamic tasks of different difficulty levels.
Remote monitoring of physical activity | over 7 days at 1 week before TKA, 7 days during the 12th , 24th and 52th week after
  Participants' physical activity will be measured by a wearable sensor. accelerometer. The participant will wear ActiGraph on the right hip, near the iliac crest for 7 days except during sleeping, showering or bathing. Data from the vertical axis will be recorded in 15s epochs and be initialized using the normal filter. The data be classified into different activity levels by ActiLife V6.11.0: sedentary (0-99 counts/minute), light (100-2019 counts/minute), moderate (2020-5998 counts/minute), and vigorous (> 5999 counts/minute).

CONTACTS AND LOCATIONS:
Overall Officials: Arnold Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University, Department of Rehabilitation Sciences
Locations (1):
- The Hong Kong Polytechnic Univeristy, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lo CWT, Brodie MA, Tsang WWN, Yan CH, Lam PL, Chan CM, Lord SR, Wong AYL. Acceptability and feasibility of a community-based strength, balance, and Tai Chi rehabilitation program in improving physical function and balance of patients after total knee arthroplasty: study protocol for a pilot randomized controlled trial. Trials. 2021 Feb 11;22(1):129. doi: 10.1186/s13063-021-05055-5. PMID 33573664